CLINICAL TRIAL: NCT00191386
Title: Long-Term Extension, Open-Label Study of Atomoxetine Hydrochloride in Child Outpatients With Attention-Deficit/Hyperactivity Disorder
Brief Title: Long-Term Study of Atomoxetine in Children With Attention-Deficit/Hyperactivity Disorder (AD/HD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9315; B4Z-JE-LYDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Experimental): 0.5 milligrams per kilogram (mg/kg) twice daily (BID), orally (PO) titrated to 1.2 mg/kg BID, PO over 2 weeks then 1.2 to 1.8 mg/kg BID, PO for 6 months and up to 4 years
  Interventions: Drug: Atomoxetine hydrochloride

INTERVENTIONS:
Drug: Atomoxetine hydrochloride — 0.5 milligrams per kilogram (mg/kg) twice daily (BID), orally (PO) titrated to 1.2 mg/kg BID, PO over 2 weeks then 1.2 to 1.8 mg/kg BID, PO for 6 months and up to 4 years
  Other Names: LY139603; Strattera

SUMMARY:
The study is long-term extension study to evaluate long-term safety and efficacy of Atomoxetine in Japanese pediatric patients with Attention-Deficit/Hyperactivity Disorder (AD/HD).

ELIGIBILITY:
Inclusion Criteria:

* Patients who met all of the disease diagnostic and study criteria at Visit 2 of previous placebo-controlled study, completed the study
* Patients wish to enter into this study

Exclusion Criteria:

* Patients whose families anticipate a move outside the geographic range of the investigative site, or who plan extended travel inconsistent with the recommended visit interval

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2005-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- Japan (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wakayama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This ongoing study is being conducted as a follow-up investigation of ADHD pediatric patients who completed Study LYBC (NCT00191295).
Period: Overall Study
Arm/Group | Atomoxetine
Started | 228
6 Months | 183
12 Months | 149
2 Years | 105
3 Years | 65
Completed | 68
Not Completed | 160
Not completed — Adverse Event | 16
Not completed — Lost to Follow-up | 1
Not completed — Entry Criteria Exclusion | 3
Not completed — Protocol Violation | 18
Not completed — Withdrawal by Subject | 96
Not completed — Physician Decision | 11
Not completed — Lack of Efficacy | 15

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
Age Continuous [Mean (Standard Deviation); unit: years] | 10.69 (2.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 195
Race/Ethnicity, Customized [Number; unit: Participants]
  East Asian | 228
Region of Enrollment [Number; unit: participants]
  Japan | 228
ADHD Rating Scale-IV-Translated in Japanese Parent Version: Investigator Administered/Scored [Mean (Standard Deviation); unit: Units on a scale] — Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD). Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
  Units on a scale | 22.23 (10.42)
Clinical Global Impressions-Attention Deficit Hyperactivity Disorder-Severity (CGI-ADHD-S) [Mean (Standard Deviation); unit: Units on a scale] — Measures total improvement (or worsening) of a participant's ADHD symptoms from the beginning of treatment. (1=very much improved, 7=very much worsened).
  Units on a scale | 4.00 (1.04)
Mean Age at Onset of Attention Deficit Hyperactivity Disorder (ADHD) [Mean (Standard Deviation); unit: Years] | 3.93 (1.57)
Age at Onset of ADHD [Number; unit: Participants]
  0 Years | 1
  1 Years | 17
  2 Years | 25
  3 Years | 49
  4 Years | 45
  5 Years | 47
  6 Years | 40
  7 Years | 4
Duration of ADHD [Mean (Standard Deviation); unit: Years] | 6.25 (2.85)
Duration of ADHD [Number; unit: Participants]
  1 Years | 6
  2 Years | 8
  3 Years | 30
  4 Years | 24
  5 Years | 32
  6 Years | 26
  7 Years | 31
  8 Years | 21
  9 Years | 22
  10 Years | 11
  11 Years | 4
  12 Years | 7
  13 Years | 3
  14 Years | 3
Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-PL [Number; unit: Participants with Disorder Presently] — The Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime Version (K-SADS-PL) is a semi-structured interview schedule for assessing psychiatric disorders in children and adolescents. It is used to assess the status of 32 DSM-IV child and adolescent psychiatric diagnosis.
  Participants with Disorder Presently
    Oppositional Defiant Disorder | 32
    Conduct Disorder | 2
    Specific Phobia | 3
    Generalized Anxiety Disorder | 1
    Obsessive Compulsive Disorder | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events for Long Term Safety and Tolerability
Description: Details on the actual adverse events are presented in the Reported Adverse Events Section.
Time Frame: Baseline through 4 years
Population: All patients who took at least one dose of study medication were included in the analyses of safety data.
Measure: Number; unit: Participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
Participants
  Serious Adverse Events | 6
  All Other Nonserious Adverse Events | 222

2. Secondary Outcome: Change From Baseline at Various Timepoints in Attention Deficit Hyperactivity Disorder Rating Scale-IV-Translated in Japanese Parent Version: Investigator Administered and Scored (ADHDRS-IV-J:I) Total Score
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
Time Frame: Baseline, 6 Months, 12 Months, 2 Years, 3 Years, 4 Years
Population: Full Analysis Set: Participants who met Study LYBC criteria, took 1 dose of drug, had a baseline/post-baseline measurement. Changes from baseline used LOCF approach. Baseline was the last non-missing measurement before taking atomoxetine (either LYDA Week 0 or LYBC Week 2). Endpoint was the last non-missing measurement in each assessment period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
Units on a scale
  Total Score 6 Months (n=228) | -14.1 (9.3)
  Total Score 12 Months (n=178) | -16.0 (9.2)
  Total Score 2 Years (n=143) | -17.7 (9.4)
  Total Score 3 Years (n=105) | -20.0 (9.2)
  Total Score 4 Years (n=62) | -20.1 (10.5)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for Total Score 6 Months
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for Total Score 12 Months
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for Total Score 2 Years
Statistical Analysis 4: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for Total Score 3 Years
Statistical Analysis 5: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for Total Score 4 Years

3. Secondary Outcome: Change From Baseline at Various Timepoints in the Clinical Global Impressions-Attention Deficit Hyperactivity Disorder-Severity (CGI-ADHD-S)
Description: Measures severity of the participant's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline, 6 Months, 12 Months, 2 Years, 3 Years, 4 Years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
Units on a scale
  6 Months | -1.1 (1.1)
  12 Months | -1.3 (1.1)
  2 Years | -1.4 (1.0)
  3 Years | -1.6 (1.0)
  4 Years | -1.8 (1.1)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for 6 Months
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for 12 Months
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for 2 Years
Statistical Analysis 4: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for 3 Years
Statistical Analysis 5: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-Value for 4 Years

4. Secondary Outcome: Cytochrome P450 2D6 (CYP2D6) Phenotype Status
Description: Participants were categorized as either extensive metabolizers (EM) or poor metabolizers (PM). CYP2D6 is the primary atomoxetine metabolizing enzyme. The CYP2D6 genotype were analysed by testing the *2, *3, *4, *5, *6, *7, *8, and *10 alleles. Metabolizer status was determined by focusing on the normal(wild type, *2), decreased(*10), and defective allele(*3, *4, *5, *6, *7, or *8). PM were assigned to the patients had two defective alleles in any combination of *3, *4, *5, *6, *7, or *8 alleles. EM was all except for PM.
Time Frame: Over 1 year
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
Participants
  Extensive Metabolizer | 225
  Poor Metabolizer | 3

ADVERSE EVENTS:
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 6/228
Other Adverse Events (participants affected / at risk) | 222/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=228)
Thyroiditis (Endocrine disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=228)
Conjunctivitis allergic (Eye disorders) | 13 (17)
Myopia (Eye disorders) | 12 (13)
Abdominal pain (Gastrointestinal disorders) | 53 (106)
Constipation (Gastrointestinal disorders) | 17 (25)
Dental caries (Gastrointestinal disorders) | 23 (24)
Diarrhoea (Gastrointestinal disorders) | 42 (58)
Nausea (Gastrointestinal disorders) | 28 (47)
Stomatitis (Gastrointestinal disorders) | 20 (27)
Toothache (Gastrointestinal disorders) | 12 (12)
Vomiting (Gastrointestinal disorders) | 29 (45)
Malaise (General disorders) | 14 (20)
Pyrexia (General disorders) | 34 (43)
Bronchitis (Infections and infestations) | 23 (39)
Gastroenteritis (Infections and infestations) | 36 (53)
Gastroenteritis viral (Infections and infestations) | 18 (25)
Impetigo (Infections and infestations) | 15 (17)
Influenza (Infections and infestations) | 55 (62)
Nasopharyngitis (Infections and infestations) | 127 (420)
Otitis media (Infections and infestations) | 12 (14)
Pharyngitis (Infections and infestations) | 26 (46)
Rhinitis (Infections and infestations) | 17 (31)
Arthropod sting (Injury, poisoning and procedural complications) | 18 (41)
Contusion (Injury, poisoning and procedural complications) | 30 (51)
Excoriation (Injury, poisoning and procedural complications) | 17 (30)
Fall (Injury, poisoning and procedural complications) | 18 (26)
Joint sprain (Injury, poisoning and procedural complications) | 22 (30)
Decreased appetite (Metabolism and nutrition disorders) | 30 (36)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (17)
Headache (Nervous system disorders) | 67 (173)
Somnolence (Nervous system disorders) | 34 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 (55)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 22 (30)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 49 (139)
Eczema (Skin and subcutaneous tissue disorders) | 21 (29)
Urticaria (Skin and subcutaneous tissue disorders) | 12 (24)
Tooth extraction (Surgical and medical procedures) | 14 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days